CLINICAL TRIAL: NCT00000133
Title: Cryotherapy for Retinopathy of Prematurity (CRYO-ROP) - Outcome Study of Cryotherapy for Retinopathy of Prematurity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Allocation: Randomized
Other Study IDs: NEI-32
Record Dates: First submitted 1999-09-23; First posted 1999-09-24 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2003-10

CONDITIONS: Retinopathy of Prematurity
MeSH Terms: conditions — Retinopathy of Prematurity

INTERVENTIONS:
Procedure: Trans-scleral Cryotherapy

SUMMARY:
To determine the safety and efficacy of trans-scleral cryotherapy of the peripheral retina in certain low birth-weight infants with retinopathy of prematurity (ROP) for reducing blindness from ROP.

To determine the long-term outcome for eyes that had severe ("threshold") ROP, both with and without cryotherapy.

DETAILED DESCRIPTION:
ROP is a disease of the eyes of prematurely born infants in which the retinal blood vessels increase in number and branch excessively, sometimes leading to hemorrhage or scarring. Before the establishment of this study in 1985, more than 500 infants annually were blinded by ROP in the United States alone.

More than 30 years ago, the National Institutes of Health sponsored a clinical trial that showed that if premature babies are given oxygen only as needed, the number of infants who develop ROP drops dramatically. Subsequently, hospitals cut back on giving excessive oxygen routinely to premature babies. But, with improvements in neonatal care over the last two decades, the number of babies at risk is increasing as survival rates for smaller premature infants improve. The lower the birth weight, the higher the incidence and severity of ROP.

In a more recent NEI-supported study at the University of Miami, blood oxygen levels of very low birth-weight infants were monitored continuously by use of transcutaneous measurements as long as oxygen therapy was needed. The study showed that there is no statistically significant difference between the rates of ROP in infants monitored on continuous oxygen therapy and in those monitored only when they were receiving oxygen in excess of 40 percent.

The Supplemental Therapeutic Oxygen for Prethreshold ROP (STOP-ROP) trial, also funded by the NEI, studied whether a slight increase in oxygen therapy would prevent the progression of moderate ROP to ROP severe enough to require surgical treatment. This intervention made little or no difference in outcomes.

Likewise, another NEI-sponsored clinical trial (LIGHT-ROP) demonstrated absence of protective effect on ROP by limiting light exposure to newborn premature infants. These studies have led to the conclusion that factors other than oxygen or light exposure must be involved in causing ROP.

In most infants who develop ROP, the disease spontaneously subsides, permitting development of normal vision. But other infants who progress to a severe form of ROP are in danger of becoming permanently blind. Although the cause of ROP is not fully explained, scientists are seeking ways to treat ROP successfully and to find the right time in the progression of the disease to use treatment. Cryotherapy, which destroys the fringe of the retina through freezing, is the only treatment so far that has been demonstrated to provide substantial benefit to these eyes.

The multicenter trial of cryotherapy for ROP enrolled more than 4,000 premature infants who weighed no more than 1,250 grams at birth. This category of infants is at the greatest risk of developing ROP. The eyes of the infants enrolled in the study were examined at predetermined intervals while the subjects were still in the intensive care nursery. After the pupils were dilated with eye drops, the eyes were examined by an ophthalmologist using a binocular indirect ophthalmoscope to visualize the developing retina. The natural history of the condition of each infant's retina was recorded. When examination disclosed the severe form of ROP (threshold ROP) in both eyes, and the parents gave informed consent, one of the infant's eyes was randomly selected to receive cryotherapy. In this technique, a cryoprobe was used to freeze and thus destroy the peripheral extent of the retina, thereby arresting the development of the blood vessels growing wildly toward it.

Outcome of the therapy was assessed at 3 months and 12 months following randomization by an extensive examination that included photography of the interior of both the treated and the control eyes. The 12-month exam also measured visual function with preferential-looking techniques. Such measurements allowed correlations between fundus photographs and visual function and a comparison of visual function for treated versus control eyes. Neither the trained photograph readers who evaluated the pictures from both eyes nor the specially trained vision testers knew which eyes had received cryotherapy. Additional assessments of visual acuity and retinal status have been made approximately each year up to the present. Currently (2001), preparations are being made for a 15-year outcome study that will conclude by 2003.

ELIGIBILITY:
Premature infants of either gender who were eligible for the natural history study had weighed less than 1,251 grams at birth and had survived the first 28 days of life. They had no major ocular or systemic congenital anomalies. Infants who met these criteria and also had a threshold level of ROP (defined as stage 3+ of the International Classification of Retinopathy of Prematurity occupying five or more contiguous or eight cumulative 30 degree sectors [clock hours] of stage 3 ROP in zone I or II in the presence of plus disease) could be referred for examination to determine eligibility for entry to the cryotherapy trial.

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 1986-01; Study Completion 2003-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - Alabama Ophthalmology Associates, P.C., Birmingham, Alabama
  - Private practice of David Plotsky, MD, Washington D.C., District of Columbia
  - Retina Group of Washington, Washington D.C., District of Columbia
  - Bascom Palmer Eye Institute, University of Miami School of Medicine, Miami, Florida
  - University of Illinois Eye and Ear Infirmary, Chicago, Illinois
  - Department of Ophthalmology, Indiana University School of Medicine, Indianapolis, Indiana
  - Kentucky Lions Eye Research Institute, University of Louisville, Louisville, Kentucky
  - Department of Ophthalmology, Tulane University School of Medicine, New Orleans, Louisiana
  - Wilmer Eye Institute, The Johns Hopkins Medical Institutions, Baltimore, Maryland
  - Private practice of John D. Baker, MD, Dearborn, Michigan
  - Associated Retinal Consultants, P.C., Royal Oak, Michigan
  - Department of Ophthalmology, University of Minnesota, Minneapolis, Minnesota
  - Strong Children's Hospital, University of Rochester Medical Center, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Private Practice of Miles J. Burke, MD, Cincinnati, Ohio
  - Columbus Children's Hospital, Columbus, Ohio
  - Oregon Health & Science University, Casey Eye Institute, Portland, Oregon
  - Children's Hospital of Philadelphia, Division of Pediatric Ophthalmology, Philadelphia, Pennsylvania
  - Pediatric Ophthalmology and Strabismus, Inc., Pittsburgh, Pennsylvania
  - Storm Eye Institute, Medical University of South Carolina, Charleston, South Carolina
  - Department of Ophthalmology, Vanderbilt University Medical Center, Nashville, Tennessee
  - Private practice of Rand Spencer, M.D., Dallas, Texas
  - University of Texas Health Science Center, San Antonio, Department of Ophthalmology, San Antonio, Texas
  - John Moran Eye Center, Salt Lake City, Utah

REFERENCES:
- [Background] Multicenter trial of cryotherapy for retinopathy of prematurity: preliminary results. Cryotherapy for Retinopathy of Prematurity Cooperative Group. Pediatrics. 1988 May;81(5):697-706. PMID 2895910
- [Background] Multicenter trial of cryotherapy for retinopathy of prematurity. Three-month outcome. Cryotherapy for Retinopathy of Prematurity Cooperative Group. Arch Ophthalmol. 1990 Feb;108(2):195-204. doi: 10.1001/archopht.1990.01070040047029. PMID 2405827
- [Background] Dobson V, Quinn GE, Biglan AW, Tung B, Flynn JT, Palmer EA. Acuity card assessment of visual function in the cryotherapy for retinopathy of prematurity trial. Invest Ophthalmol Vis Sci. 1990 Sep;31(9):1702-8. PMID 2211019
- [Background] Watzke RC, Robertson JE Jr, Palmer EA, Wallace PR, Evans MS, Soldevilla JE. Photographic grading in the retinopathy of prematurity cryotherapy trial. Arch Ophthalmol. 1990 Jul;108(7):950-5. doi: 10.1001/archopht.1990.01070090052038. PMID 2369354
- [Background] Hardy RJ, Davis BR, Palmer EA, Tung B. Statistical considerations in terminating randomization in the Multicenter Trial of Cryotherapy for Retinopathy of Prematurity. Cryotherapy for Retinopathy of Prematurity Cooperative Group. Control Clin Trials. 1991 Apr;12(2):293-303. doi: 10.1016/0197-2456(91)90026-i. PMID 1645641
- [Background] Palmer EA, Flynn JT, Hardy RJ, Phelps DL, Phillips CL, Schaffer DB, Tung B. Incidence and early course of retinopathy of prematurity. The Cryotherapy for Retinopathy of Prematurity Cooperative Group. Ophthalmology. 1991 Nov;98(11):1628-40. doi: 10.1016/s0161-6420(91)32074-8. PMID 1800923
- [Background] Palmer EA, Hardy RJ, Davis BR, Stein JA, Mowery RL, Tung B, Phelps DL, Schaffer DB, Flynn JT, Phillips CL. Operational aspects of terminating randomization in the Multicenter Trial of Cryotherapy for Retinopathy of Prematurity. Cryotherapy for Retinopathy of Prematurity Cooperative Group. Control Clin Trials. 1991 Apr;12(2):277-92. doi: 10.1016/0197-2456(91)90025-h. PMID 1645640
- [Background] Phelps DL, Brown DR, Tung B, Cassady G, McClead RE, Purohit DM, Palmer EA. 28-day survival rates of 6676 neonates with birth weights of 1250 grams or less. Pediatrics. 1991 Jan;87(1):7-17. PMID 1984621
- [Background] Quinn GE, Dobson V, Barr CC, Davis BR, Flynn JT, Palmer EA, Robertson J, Trese MT. Visual acuity in infants after vitrectomy for severe retinopathy of prematurity. Ophthalmology. 1991 Jan;98(1):5-13. doi: 10.1016/s0161-6420(91)32343-1. PMID 2023732
- [Background] Gilbert WS, Dobson V, Quinn GE, Reynolds J, Tung B, Flynn JT. The correlation of visual function with posterior retinal structure in severe retinopathy of prematurity. Cryotherapy for Retinopathy of Prematurity Cooperative Group. Arch Ophthalmol. 1992 May;110(5):625-31. doi: 10.1001/archopht.1992.01080170047022. PMID 1580837
- [Background] Quinn GE, Dobson V, Repka MX, Reynolds J, Kivlin J, Davis B, Buckley E, Flynn JT, Palmer EA. Development of myopia in infants with birth weights less than 1251 grams. The Cryotherapy for Retinopathy of Prematurity Cooperative Group. Ophthalmology. 1992 Mar;99(3):329-40. doi: 10.1016/s0161-6420(92)31968-2. PMID 1565444
- [Background] Summers G, Phelps DL, Tung B, Palmer EA. Ocular cosmesis in retinopathy of prematurity. The Cryotherapy for Retinopathy of Prematurity Cooperative Group. Arch Ophthalmol. 1992 Aug;110(8):1092-7. doi: 10.1001/archopht.1992.01080200072027. PMID 1497522
- [Background] Trueb L; Evans J; Hammel A; Bartholomew P; Dobson D; Assessing visual acuity of visually impaired children using the Teller acuity cards., Am Orthoptic J 1992;42:149-154
- [Background] Multicenter trial of cryotherapy for retinopathy of prematurity. 3 1/2-year outcome--structure and function. Cryotherapy for Retinopathy of Prematurity Cooperative Group. Arch Ophthalmol. 1993 Mar;111(3):339-44. PMID 8447743
- [Background] Evans MS; Wallace PR; Palmer EA; Fundus photography in small infants., J Ophthal Photography 1993;15(1):38-39
- [Background] Reynolds J, Dobson V, Quinn GE, Gilbert WS, Tung B, Robertson J, Flynn JT. Prediction of visual function in eyes with mild to moderate posterior pole residua of retinopathy of prematurity. Cryotherapy for Retinopathy of Prematurity Cooperative Group. Arch Ophthalmol. 1993 Aug;111(8):1050-6. doi: 10.1001/archopht.1993.01090080046017. PMID 8352687
- [Background] Schaffer DB, Palmer EA, Plotsky DF, Metz HS, Flynn JT, Tung B, Hardy RJ. Prognostic factors in the natural course of retinopathy of prematurity. The Cryotherapy for Retinopathy of Prematurity Cooperative Group. Ophthalmology. 1993 Feb;100(2):230-7. doi: 10.1016/s0161-6420(93)31665-9. PMID 8437832
- [Background] The natural ocular outcome of premature birth and retinopathy. Status at 1 year. Cryotherapy for Retinopathy of Prematurity Cooperative Group. Arch Ophthalmol. 1994 Jul;112(7):903-12. doi: 10.1001/archopht.1994.01090190051021. PMID 8031269
- [Background] Dobson V, Quinn GE, Summers CG, Saunders RA, Phelps DL, Tung B, Palmer EA. Effect of acute-phase retinopathy of prematurity on grating acuity development in the very low birth weight infant. The Cryotherapy for Retinopathy of Prematurity Cooperative Group. Invest Ophthalmol Vis Sci. 1994 Dec;35(13):4236-44. PMID 8002243
- [Background] Dobson V, Quinn GE, Saunders RA, Spencer R, Davis BR, Risser J, Palmer EA. Grating visual acuity in eyes with retinal residua of retinopathy of prematurity. The Cryotherapy for Retinopathy of Prematurity Cooperative Group. Arch Ophthalmol. 1995 Sep;113(9):1172-7. doi: 10.1001/archopht.1995.01100090098029. PMID 7661752
- [Background] Dobson V, Quinn GE, Tung B, Palmer EA, Reynolds JD. Comparison of recognition and grating acuities in very-low-birth-weight children with and without retinal residua of retinopathy of prematurity. Cryotherapy for Retinopathy of Prematurity Cooperative Group. Invest Ophthalmol Vis Sci. 1995 Mar;36(3):692-702. PMID 7890499
- [Background] Kivlin JD, Biglan AW, Gordon RA, Dobson V, Hardy RA, Palmer EA, Tung B, Gilbert W, Spencer R, Cheng KP, Buckley E. Early retinal vessel development and iris vessel dilatation as factors in retinopathy of prematurity. Cryotherapy for Retinopathy of Prematurity (CRYO-ROP) Cooperative Group. Arch Ophthalmol. 1996 Feb;114(2):150-4. doi: 10.1001/archopht.1996.01100130144005. PMID 8573016
- [Background] Quinn GE, Dobson V, Biglan A, Evans J, Plotsky D, Hardy RJ. Correlation of retinopathy of prematurity in fellow eyes in the cryotherapy for retinopathy of prematurity study. The Cryotherapy for Retinopathy of Prematurity Cooperative Group. Arch Ophthalmol. 1995 Apr;113(4):469-73. doi: 10.1001/archopht.1995.01100040089032. PMID 7710397
- [Background] Bartholomew PA; Chao J; Evans JL; Hammel AM; Trueb AL; Verness JL; Dobson V; Quinn GE; Acceptance/Use of the Teller acuity card procedure in the clinic., Am Orthoptic J 1996;46:100-106
- [Background] Cryotherapy for Retinopathy of Prematurity Cooperative Group. Multicenter trial of cryotherapy for retinopathy of prematurity. Snellen visual acuity and structural outcome at 5 1/2 years after randomization. Arch Ophthalmol. 1996 Apr;114(4):417-24. doi: 10.1001/archopht.1996.01100130413008. PMID 8602778
- [Background] Dobson V, Quinn GE, Abramov I, Hardy RJ, Tung B, Siatkowski RM, Phelps DL. Color vision measured with pseudoisochromatic plates at five-and-a-half years in eyes of children from the CRYO-ROP study. Invest Ophthalmol Vis Sci. 1996 Nov;37(12):2467-74. PMID 8933763
- [Background] Gilbert WS, Quinn GE, Dobson V, Reynolds J, Hardy RJ, Palmer EA. Partial retinal detachment at 3 months after threshold retinopathy of prematurity. Long-term structural and functional outcome. Multicenter Trial of Cryotherapy for Retinopathy of Prematurity Cooperative Group. Arch Ophthalmol. 1996 Sep;114(9):1085-91. doi: 10.1001/archopht.1996.01100140287005. PMID 8790093
- [Background] Quinn GE, Dobson V, Barr CC, Davis BR, Palmer EA, Robertson J, Summers CG, Trese MT, Tung B. Visual acuity of eyes after vitrectomy for retinopathy of prematurity: follow-up at 5 1/2 years. The Cryotherapy for Retinopathy of Prematurity Cooperative Group. Ophthalmology. 1996 Apr;103(4):595-600. doi: 10.1016/s0161-6420(96)30647-7. PMID 8618758
- [Background] Quinn GE, Dobson V, Hardy RJ, Tung B, Phelps DL, Palmer EA. Visual fields measured with double-arc perimetry in eyes with threshold retinopathy of prematurity from the cryotherapy for retinopathy of prematurity trial. The CRYO-Retinopathy of Prematurity Cooperative Group. Ophthalmology. 1996 Sep;103(9):1432-7. doi: 10.1016/s0161-6420(96)30487-9. PMID 8841302
- [Background] Hardy RJ, Palmer EA, Schaffer DB, Phelps DL, Davis BR, Cooper CJ. Outcome-based management of retinopathy of prematurity. Multicenter Trial of Cryotherapy for Retinopathy of prematurity Cooperative Group. J AAPOS. 1997 Mar;1(1):46-54. doi: 10.1016/s1091-8531(97)90023-9. PMID 10530985
- [Background] Saunders RA, Donahue ML, Christmann LM, Pakalnis AV, Tung B, Hardy RJ, Phelps DL. Racial variation in retinopathy of prematurity. The Cryotherapy for Retinopathy of Prematurity Cooperative Group. Arch Ophthalmol. 1997 May;115(5):604-8. doi: 10.1001/archopht.1997.01100150606005. PMID 9152127
- [Background] Multicenter trial of cryotherapy for retinopathy of prematurity. Preliminary results. Cryotherapy for Retinopathy of Prematurity Cooperative Group. Arch Ophthalmol. 1988 Apr;106(4):471-9. doi: 10.1001/archopht.1988.01060130517027. PMID 2895630